CLINICAL TRIAL: NCT06959810
Title: Impact of Adapted Aesthetic Onco in Patients With Cancer of the Upper Aero-digestive Tract During Their Management [ŒUVRE (Adapted Aesthetic Onco Aero-digestive Tract)]
Brief Title: Impact of Adapted Aesthetic Onco in Patients With Upper Aerodigestive Tract Cancer During Their Management
Acronym: OEUVRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Fondation de France (Other); GIRCI NO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OEUVRE
Record Dates: First submitted 2025-04-23; First posted 2025-05-07 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Oncology; Aerodigestive Tract Cancer; Suportive Care
Keywords: Oncology (Organ: Upper Aero Digestive Tract); Supportive Oncology; Organization of care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three sessions of Adapted Onco-Esthetics (Experimental): Patients will received three sessions of Adapted Onco-Esthetics
  Interventions: Other: Adapted Onco-Esthetics sessions

INTERVENTIONS:
Other: Adapted Onco-Esthetics sessions — Patient will received three sessions of Adapted Onco-Esthetics

SUMMARY:
Treatment for cancers of the pharyngolarynx is mutilating, with major consequences for patients' lives in terms of physical and functional after-effects. The psycho-social consequences are also significant, notably the metamorphosis of identity linked to the disease and its treatment, which alters the patient's self-image.

Initial feedback from patients who have been able to benefit from adapted oncoesthetics (OEA) is overwhelmingly positive.

This study will assess the feasibility of oncoesthetics and describe any obstacles.

DETAILED DESCRIPTION:
The majority of patients treated for VADS cancer come from disadvantaged socio-professional and family backgrounds. Treatment for cancers of the pharyngolarynx is mutilating, with major consequences for patients' lives in terms of physical and functional after-effects. The psycho-social consequences are also significant, notably the metamorphosis of identity linked to the disease and its treatment, which alters the patient's self-image.

The French association for Oncological Support Care (SOS) defines socio-aesthetics as "the professional practice of aesthetic care adapted to people who are fragile or suffering as a result of an attack on their physical or psychological integrity, or in social distress". Priority patients for aesthetic care are those whose treatments have had an impact on body image (mutilating surgery, skin toxicities), and/or who are in a situation of social precariousness and suffer from a loss of self-esteem.

For patients suffering from VADS cancer, a population not usually in need of aesthetic care but in need of self-image restoration, an incentive program has been set up. Initial feedback from patients who have been able to benefit from adapted oncoesthetics (OEA) is overwhelmingly positive.

This study will assess the feasibility of OAS for VADS cancer patients, and describe any obstacles.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Neoplastic location: oropharynx, oral cavity, hypopharynx, larynx, nasal cavity, salivary glands, cavum, sinus.
* Patient due to start oncological treatment (recurrence authorized)
* Patient fluent in French.
* Affiliation with a social security scheme
* Signature of informed consent prior to any specific procedure linked to the study
* Treatment with curative intent

Exclusion Criteria:

* Breast-feeding or pregnant patient
* Any associated medical or psychological condition that could compromise the patient's ability to participate in the study
* Patient deprived of liberty, under guardianship, or subject to a legal protection measure or unable to express their consent.
* Patient unable to undergo trial follow-up for geographical, social or psychopathological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-09-16 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate, in patients treated for cancer of the upper aerodigestive tract, the impact of early treatment with Adapted Onco-Esthetics | At each session (first , second and third). An interval of one to 4 weeks between 2 sessions is permitted
  Evaluation of the proportion of patients reporting no worsening of self-image representation, as measured by the BIS body image scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Francois Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: No